CLINICAL TRIAL: NCT02128893
Title: A Phase 1 Randomized Open Label, Parallel Group Study to Evaluate the Effect of Multiple Doses of Esomeprazole on the Pharmacokinetics of Isavuconazole
Brief Title: A Study to Evaluate the Effect of Multiple Doses of Esomeprazole on the Pharmacokinetics of Isavuconazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Basilea Pharmaceutica International Ltd (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 9766-CL-0054
Record Dates: First submitted 2014-04-30; First posted 2014-05-01 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Pharmacokinetics of Isavuconazole; Healthy Subjects
Keywords: Isavuconazole; Esomeprazole; BAL4815; BAL8728; Healthy Subjects
MeSH Terms: interventions — isavuconazole; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isavuconazole alone (Experimental): Isavuconazole three times a day on Days 1 and 2 and once a day on Days 3, 4, and 5
  Interventions: Drug: Isavuconazole
- Isavuconazole and Esomeprazole (Experimental): Esomeprazole daily for 10 days starting on Day 1 and isavuconazole three times a day on Days 6 and 7 and once a day on Days 8, 9, and 10
  Interventions: Drug: Isavuconazole; Drug: Esomeprazole

INTERVENTIONS:
Drug: Isavuconazole — oral
  Other Names: BAL4815
Drug: Esomeprazole — oral
  Other Names: Nexium®
  Arms: Isavuconazole and Esomeprazole

SUMMARY:
The purpose of this study is to assess the effect of multiple doses of esomeprazole on the pharmacokinetics of isavuconazole. In addition, safety and tolerability of isavuconazole alone and in combination with esomeprazole will be assessed

ELIGIBILITY:
Inclusion Criteria:

* The subject has a body weight of at least 50 kg and a body mass index of 18.5 to 32 kg/m2, inclusive
* The subject's 12-lead electrocardiogram (ECG) is normal
* The subject's clinical laboratory test results are within normal limits

Exclusion Criteria:

* The subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy
* The subject has a history of bowel obstruction, swallowing disorder, severe gastro-intestinal disorders, major gastrointestinal surgery, gastric/duodenal ulcers or any other condition that may interfere with study drug absorption
* Female subject has been pregnant within 6 months before screening or breast feeding within 3 months before screening
* The subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmia or torsade de pointes, structural heart disease, or family history of either Short or Long QT syndrome (suggested by sudden death of a close relative at a young age due to possible or probable cardiac causes). QT is the time between the start of the Q wave and the end of the T wave in the heart's electrical system
* The subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to clinic admission
* The subject has received a vaccination within the last 30 days prior to study drug administration
* The subject has a positive serology test for Hepatitis B surface antigen (HBsAg), Hepatitis A Immunoglobulin M antibody (anti HAV (IgM)), Hepatitis C antibody (anti-HCV), or human immunodeficiency virus (anti-HIV 1+2)
* The subject has a known or suspected allergy to any of the components of the trial products or the azole class of compounds, or a history of multiple and/or severe allergies to drugs or foods, or a history of severe anaphylactic reactions
* The subject has used tobacco or nicotine containing products in the last 6 months
* The subject has had treatment with any prescribed or non-prescribed drugs (including vitamins, natural and herbal remedies, e.g. St. John's wort) in the 2 weeks prior with the exception of hormonal methods of contraception, hormone replacement therapy, or occasional use of acetaminophen up to 2 g/day
* The subject has participated in any interventional clinical study or has received any investigational drugs within past 30 days or 5 half-lives, whichever is longer
* The subject has had any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to clinic admission
* The subject anticipates an inability to abstain from alcohol or caffeine use for 48 hours prior and throughout the duration of the study; or from grapefruit, grapefruit juice, star fruit, or Seville oranges or any products containing these items from 72 hours prior and throughout the duration of the study
* The subject has history of consuming more than 14 units of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical/substance abuse within past 2 years prior to screening (Note: one unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits/hard liquor) or the subject tests positive for alcohol or drugs of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, and opiates)
* The subject has taken part in strenuous exercise within 3 days before Day 1

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of plasma isavuconazole concentration: Area under the concentration-time curve during the time interval between consecutive dosing (AUCtau) | Day 5 (Arm 1) and Day 10 (Arm 2)
Pharmacokinetics of plasma isavuconazole concentration: Maximum concentration (Cmax) | Day 5 (Arm 1) and Day 10 (Arm 2)
Pharmacokinetics of plasma isavuconazole concentration: Time after dosing when Cmax occurs (tmax) | Day 5 (Arm 1) and Day 10 (Arm 2)
Safety assessed through adverse events | up to Day 17
Safety assessed through clinical laboratory evaluations | up to Day 11
  Laboratory assessments will include hematology, serum chemistry and urinalysis parameters
Safety assessed by 12-lead electrocardiograms (ECGs) | up to Day 11
Safety assessed through vital signs | up to Day 11
  Vital signs will be measured including oral temperature, pulse, and sitting blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (1):
- Parexel Early Phase Clinical Unit, Baltimore, Maryland, United States